CLINICAL TRIAL: NCT04701320
Title: Clinical Evaluation of Nano Hydroxyapatite Reinforced Glass Ionomer Versus Conventional Glass Ionomer in Treatment of Root Caries in Geriatric Patients: A Randomized Controlled Clinical Trial
Brief Title: Clinical Evaluation of Nano Hydroxyapatite Reinforced Glass Ionomer in Treatment of Root Caries in Geriatric Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reham nabil mahmoud, associate lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OPER 3-3-6
Record Dates: First submitted 2020-07-25; First posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Dental Restoration Failure
Keywords: Glass Carbomer GCP glass fill root caries Clinical perfomance
MeSH Terms: interventions — glass carbomer cement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glass carbomer (Experimental): Nano hydroxyapatite Reinforced Glass Ionomer that results in chemical bond formation with tooth structure mimic that of enamel tissue
  Interventions: Drug: Nano hydroxyapatite reinforced glass ionomer
- Fuji ix (Active Comparator): Conventional Glass Ionomer cement fluoride-releasing restorative system that combines fluoride release of glass ionomer cement and acceptable esthetics, a wear resistant, self-adhesive
  Interventions: Drug: Conventional glass ionomer

INTERVENTIONS:
Drug: Conventional glass ionomer — Conventional glass ionomer with enhanced mechanical and esthetic proberties
  Other Names: Fujiix gc corporation
  Arms: Fuji ix
Drug: Nano hydroxyapatite reinforced glass ionomer — Nanohydroxyapatite reinforced glass ionomer restorative material with enhanced mechanical proberties and chemical adhesion to tooth structure
  Other Names: Glass carbomer
  Arms: Glass carbomer

SUMMARY:
In geriatric patients, will the clinical performance of nano hydroxyapatite reinforced glass ionomer be better than conventional glass ionomer cement in treatment of root caries lesions over one year follow up?

DETAILED DESCRIPTION:
Glass carbomers are commercialized under the name of GCP Glass Fill, this material may be an interesting subject of research, certainly its bioactive properties as the manufacturer claims this material to have remineralizing properties. If this is the case, GCP Glass Fill could be an interesting reference material for further bioactivity studies

ELIGIBILITY:
Inclusion Criteria:

* • ≥ 50 years old

  * Males or females.
  * Community-dwelling
  * Have five or more of their own teeth
  * With ≥ 1 root caries lesion

Exclusion Criteria:

* • Patients younger than 50 years old

  * Disabilities.
  * Systemic diseases or severe medically compromised.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-07-07 (Actual); Primary Completion 2019-07-07 (Actual); Study Completion 2021-08-09 (Estimated)

PRIMARY OUTCOMES:
Clinical restorative performance Service (USHPS) | Change from the baseline at 3, 6 and12 months
  Change in the clinical behavior of the restoration (e.g. anatomical contour, shade match, secondary caries) using modified United State Public Health clinical evaluation assessment method Service (USHPS)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: one year